CLINICAL TRIAL: NCT02430142
Title: Microcirculatory Oxygen Uptake in Sepsis, Severe Sepsis and Septic Shock
Brief Title: Microcirculatory Oxygen Uptake in Sepsis
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Timo Sturm, Dr. med. Timo Sturm, DESA, Universitätsmedizin Mannheim
Other Study IDs: 2014-428M-MA
Record Dates: First submitted 2015-04-16; First posted 2015-04-30 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
Keywords: microcirculation; oxygen uptake; hypoxia; adenosine; central venous saturation; hypoxanthine; laserdoppler
MeSH Terms: conditions — Sepsis; Shock, Septic; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Vasoocclusive testing in sepsis: Septic patients defined according to the Surviving Sepsis Campaign (SSC)
  Interventions: Other: Vasoocclusive testing
- Vasoocclusive testing in severe sepsis: Severe septic patients defined according to the Surviving Sepsis Campaign (SSC)
  Interventions: Other: Vasoocclusive testing
- Vasoocclusive testing in sepsic shock: Septic shock patients defined according to the Surviving Sepsis Campaign (SSC)
  Interventions: Other: Vasoocclusive testing

INTERVENTIONS:
Other: Vasoocclusive testing — Forearm vasoocclusive testing with a laser-doppler spectrophotometry system, transpulmonary thermodilution and blood sampling;

SUMMARY:
Forearm vasoocclusive testing (VOT) will be performed with laser-doppler spectrophotometry system in septic patients on ICU. Microcirculatory oxygen uptake will be checked for prognostic value and for associations with tissue hypoxia markers and high central venus saturations.

DETAILED DESCRIPTION:
Sepsis remains a common entity in critical care patients with remarkable mortality. Microcirculatory dysfunction plays a pivotal role in the pathophysiology of sepsis and organ dysfunction. The main causal mechanisms are vasoactive substances such as nitric oxide and endothelin, destroyed endothelial surfaces and microvascular occlusion by activated coagulation and leucocytes. Furthermore there is some knowledge from vasooclussive testing (VOT) based on near-infrared spectroscopy (NIRS) and assessing the proportion of perfused vessels determined with orthogonal polarization spectral and sidestream darkfield imaging techniques (SDF) that impaired microcirculation is associated with organ dysfunction and increased mortality. Despite these well-recognised evidence previous trails proving therapy guidance with microcirculatory parameters failed in demonstrating optimised outcome . Recent guidelines still recommend fluid therapy based on central venous pressure, mean arterial pressure, urine output and or blood lactate concentration. But especially the parameter central venous oxygen saturation (ScvO2) seems to be not unproblematic. Retrospective data analysis found higher mortality rates if ScvO2 is elevated.

In the present study patients with sepsis, severe sepsis and septic shock will be evaluated on day 1 and day 4 and a follow up will be performed on day 180.

Additional to clinical parameters of organ function, infection markers, global parameters of tissue hypoxia will be captured by measurements of adenosine and whose metabolites.

Macrocirculatory cardiovascular function delivered by transpulmonary thermodilution technique will be assessed and local tissue perfusion and oxygen uptake will be measured with a transcutaneous laser-doppler spectrophotometry system in VOT.

The aim of this study is to check:

1. Is microcirculatory oxygen uptake a prognostic value in sepsis?
2. Is it correlated with biomarkers of hypoxia?
3. Are high levels of ScvO2 caused by microcirculatory impairments or by hyperdynamic macrocirculation?

ELIGIBILITY:
Inclusion Criteria:

* Criteria according to the SSC for sepsis, severe sepsis and septic shock
* Admission to the ICU within 24 hours

Exclusion Criteria:

* Pregnancy
* Cardiopulmonary resuscitation within the last 5 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted a surgical intensive care unit within the last 24 hours and the diagnosis of sepsis, severe sepsis and septic shock according to the Surviving Sepsis Campaign.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2015-04; Primary Completion 2016-10 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 180 days
  ICU-Mortality, 60-days-mortlity, 180-days-mortality will be recorded and correlated with baseline and postischemic microcirculatory oxygen delivery and uptake.

SECONDARY OUTCOMES:
Connection between ScvO2 and microcirculatory oxygen uptake | Day 1 and day 4
  The investigators will prove, if high values of central venous saturation (>75%) are associated with impaired tissue oxygen uptake.
Connection between adenosine-metabolites and microcirculatory oxygen uptake | Day 1 and day 4
  The investigators will prove, if high values of the adenosine-metabolite hypoxanthine (ng/ml) in plasma are associated with impaired tissue oxygen uptake.
Physical condition | 180 days
  Physical status at 180 days (Rankin-Scale) will be recorded and correlated with baseline and postischemic microcirculatory oxygen delivery and uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Thiel, Prof. Dr. med., Study Chair — Department of Anaesthesiology and Surgical Intensive Care, University Medical Centre of Mannheim
Locations (1):
- University Medical Centre, Department of Anaesthesiology and Surgical Intensive Care Medicine, Mannheim, Germany

REFERENCES:
- [Background] Angus DC, van der Poll T. Severe sepsis and septic shock. N Engl J Med. 2013 Aug 29;369(9):840-51. doi: 10.1056/NEJMra1208623. No abstract available. PMID 23984731
- [Background] De Backer D, Donadello K, Cortes DO. Monitoring the microcirculation. J Clin Monit Comput. 2012 Oct;26(5):361-6. doi: 10.1007/s10877-012-9383-8. Epub 2012 Jul 26. PMID 22833180
- [Background] Shapiro NI, Arnold R, Sherwin R, O'Connor J, Najarro G, Singh S, Lundy D, Nelson T, Trzeciak SW, Jones AE; Emergency Medicine Shock Research Network (EMShockNet). The association of near-infrared spectroscopy-derived tissue oxygenation measurements with sepsis syndromes, organ dysfunction and mortality in emergency department patients with sepsis. Crit Care. 2011;15(5):R223. doi: 10.1186/cc10463. Epub 2011 Sep 22. PMID 21939529
- [Background] Sakr Y, Dubois MJ, De Backer D, Creteur J, Vincent JL. Persistent microcirculatory alterations are associated with organ failure and death in patients with septic shock. Crit Care Med. 2004 Sep;32(9):1825-31. doi: 10.1097/01.ccm.0000138558.16257.3f. PMID 15343008
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Background] Textoris J, Fouche L, Wiramus S, Antonini F, Tho S, Martin C, Leone M. High central venous oxygen saturation in the latter stages of septic shock is associated with increased mortality. Crit Care. 2011 Jul 26;15(4):R176. doi: 10.1186/cc10325. PMID 21791065
- [Background] van der Voort PH, van Zanten M, Bosman RJ, van Stijn I, Wester JP, van Raalte R, Oudemans-van Straaten HM, Zandstra DF. Testing a conceptual model on early opening of the microcirculation in severe sepsis and septic shock: a randomised controlled pilot study. Eur J Anaesthesiol. 2015 Mar;32(3):189-98. doi: 10.1097/EJA.0000000000000126. PMID 25032942